CLINICAL TRIAL: NCT07354217
Title: Workflow Optimization During Pulse Field Ablation for Atrial Fibrillation
Acronym: PFA_workflow
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Johnson & Johnson (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 202512001MIPA
Record Dates: First submitted 2026-01-06; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Pulsed Field Ablation; Lidocaine
Keywords: Pulmonary Vein Isolation; LIDOCAINE; Pulse Field Ablation; cough suppression
MeSH Terms: interventions — Lidocaine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Aims: To evaluate the efficacy and safety of intravenous lidocaine during PFA ablation for diaphragm contraction and cough suppression.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LIDOCAINE (Experimental): Lidocaine 1 mg/kg
  Interventions: Drug: lidocaine
- Saline (Active Comparator): Saline 3~5ml
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: lidocaine — baseline SaO2, heart rate, and systolic and diastolic blood pressure will be recorded before and every 10 minutes after drug injection
  Arms: LIDOCAINE
Drug: Saline — baseline SaO2, heart rate, and systolic and diastolic blood pressure will be recorded before and every 10 minutes after drug injection
  Arms: Saline

SUMMARY:
To evaluate the efficacy and safety of intravenous lidocaine in reducing diaphragmatic contraction and suppressing the cough reflex during pulsed field ablation procedures.

DETAILED DESCRIPTION:
Atrial fibrillation is a common arrhythmia, and pulmonary vein isolation is the main treatment. The emerging pulsed field ablation (PFA) is tissue-selective and can reduce damage to adjacent organs, but it is often accompanied by phrenic nerve stimulation and cough reflex, affecting surgical stability. Intravenous lidocaine has been shown to suppress cough and hiccups, but its effect on PFA-induced responses has not been further studied. This study uses a prospective, randomized controlled trial to evaluate the effects of lidocaine on diaphragmatic contraction and cough reflex during PFA surgery, aiming to improve surgical safety and procedural smoothness.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with paroxysmal or persistent AF and are scheduled to undergo PVI.
2. Patients who can understand the study aims and protocol and are willing to follow the protocol for one year.

Exclusion Criteria:

1. Informed consent could not be obtained
2. Known allergy to study drug lidocaine.
3. Presence of thrombus in the LA or LA appendage
4. Underlying significant pulmonary disease, such as asthma or COPD needing long term maintenance therapy or documented interstitial lung disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy and safety of intravenous lidocaine during PFA ablation for diaphragm contraction and cough suppression. | 400 days
  The reduction of diaphragm contraction and dry cough frequency and intensity;
  1. the diaphragm movement distance during ablation, evaluated with intracardiac echocardiography (ICE);
  2. the cough frequency and intensity after energy application; cough frequency will be evaluated by a blinded technician, and cough intensity will be evaluated by both the technician and ICE;

SECONDARY OUTCOMES:
Acute effect (per vein) | 400DAYS
  1. the number of ablations that has to be terminated prematurely;
  2. the extra number of ablations that has to be applied to achieve entry block;
  3. the need to remap (3D electroanatomical map shifting);
Chronic effect | 400DAYS
  The AF recurrence rate within 1 year after the index procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospita, Taipei, Taiwan